CLINICAL TRIAL: NCT06019351
Title: Assessment of Mesiodistal Root Angulation Without Radiographic Guidance Versus CBCT Guidance: A Cross Sectional Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kholoud Khaled Abd ElAziz, teaching assistant, Cairo University
Other Study IDs: 711
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Mesiodistal Root Angulation - Radiographic Guidance - CBCT Guidance - Assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OrthoAnalyzer™ software — OrthoAnalyzer™ software module from 3Shape Software

SUMMARY:
Digital transformation in the orthodontic field profoundly alters the way in which orthodontic treatment is perceived and delivered, moreover it aids in creating individualized orthodontic appliances.A crucial step in digital orthodontic planning in either indirect bonding or aligner treatment is localization of mesiodistal tip. Earlier, Panoramic radiographs were formerly recommended to assist clinicians in properly identifying mesiodistal root angulation. recommended to help clinician to identify mesiodistal root angulation accurately. Owens et al. recorded clinically significant variation between the radiographic and the true root angulation. Alternatively CBCT (Cone Beam Computed Tomography) guided mesiodistal root angulation assessment has superior clinical significance compared to the routinely taken panoramic radiograph . despite its accuracy ,CBCT is not justified as a part of diagnostic records for orthodontic treatment planning following the ALARA rule . To eliminate additional x ray dose Computer aided mesiodistal root angulation identification is provided by several softwares such as OrthoAnalyzer™ ,OrthoCAD® ,and SureSmile® , however, the accuracy remains questionable. These finding may point out the importance of studying the accuracy mesiodistal identification to carry on digital workflow without the radiographic guidance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with digital models and panoramic radiograph as a routine diagnostic orthodontic record before treatment.
* Justified CBCT record taken for impacted and ectopic teeth, planning for MARPE (mini-screw assisted rapid palatal expansion)/MSE (maxillary skeletal expansion), critical tooth movements in periodontally compromised patients, surgery first cases, taken for previous studies and other reasons.

Exclusion Criteria:

* Severe crowding.
* Teeth with bizarre anatomy or severely decayed.
* Patients in mixed dentition stage.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with digital models and panoramic radiograph as a routine diagnostic orthodontic record before treatment.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-09-21 (Estimated)

PRIMARY OUTCOMES:
Outcome mesiodistal Angulation: angle between dental axis created by the software according to model clinical crown and the dental long axis guided by the CBCT. (In degrees) | through study completion, an average of 1 year".

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, El Manial, Egypt